CLINICAL TRIAL: NCT00413582
Title: Prospective Randomized Trial: Pain Management Strategy After Pectus Excavatum Repair
Brief Title: Pain Management for Pectus Excavatum Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06 08 128
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2011-12

CONDITIONS: Postoperative Pain
Keywords: Pectus Excavatum; Bar Repair; Pain Control; Pectus Excavatum Repair
MeSH Terms: conditions — Pain, Postoperative; Funnel Chest; Agnosia | interventions — Analgesia, Epidural

ARMS (2):
- 1 (Active Comparator): Epidural analgesia
  Interventions: Drug: Epidural Analgesia
- 2 (Experimental): IV narcotic analgesia
  Interventions: Drug: Patient-Controlled IV Analgesia

INTERVENTIONS:
Drug: Epidural Analgesia — Upon arrival to the operating room, patients will have a thoracic epidural (T 6-9) placed while in the sitting position. All epidural catheters will be inserted 3-5 cm within the epidural space and will be placed by attending anesthesiologists. Patients will receive midazolam 0.025 - 0.05 mg/kg IV (max 5mg) and/or fentanyl 0.5 - 2 mcg/kg IV for comfort during the procedure. Once the epidural is placed, the patient will be positioned for surgery. The epidural catheter will be initially bolused with 0.3ml/kg of ropivacaine 0.10% (max 10 ml), fentanyl 1 - 1.2 mcg/kg and clonidine 1.8 - 2mcg/kg. An infusion of ropivacaine 0.10%, fentanyl 2mcg/ml and clonidine 1.5mcg/ml will be initiated immediately at the rate of 0.3ml/kg/hr (max 10ml/hr). Intraoperatively, patients will receive intravenous fentanyl if indicated.
  Arms: 1
Drug: Patient-Controlled IV Analgesia — In the PCA arm, patients will receive fentanyl (3-6 mcg/kg) at anesthesia induction. Additional fentanyl may be administered intraoperatively as indicated. Patients who are > 35 Kg. (in keeping with current FDA approved labeling) will receive a clonidine 0.1 mg/day transdermal patch to the deltoid immediately after induction of anesthesia. Subjects in the epidural arm also receive clonidine. Upon arrival to the post anesthesia care unit, patients will be placed on a patient controlled analgesic (PCA) pump (hydromorphone: loading dose if needed; 5-6 mcg/kg continuous infusion; 5-6 mcg/kg six minute demand dose). An additional hydromorphone dose (8mcg/kg) will be available every 2 hours for pain scores of > 4/10 throughout the duration of PCA use.
  Arms: 2

SUMMARY:
The objective of this study is to scientifically evaluate two different management strategies for post-operative pain after pectus excavatum repair.

The hypothesis is that pain management without an epidural decreases hospital stay without compromising comfort.

The primary outcome variable is length of hospitalization after the intervention.

DETAILED DESCRIPTION:
This will be a single institution, prospective, randomized clinical trial involving patients who undergo the minimally invasive repair of a pectus excavatum deformity with bar placement. This is intended to be a definitive study.

Power calculations based on the known length of hospitalization listed above with α = 0.05 and power of 0.8 show the need for 55 patients in each arm. The primary end point will be reached during the hospital stay; therefore, we expect a very small amount of attrition and will intend to recruit 110. One group will undergo an attempt for epidural regional analgesia (epidural) for post-operative pain control. The other groups will receive patient controlled intravenous systemic analgesia (PCA).

Both groups will have the same management algorithm. All data will be analyzed on intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a pectus excavatum repair with bar placement.

Exclusion Criteria:

* Open repair
* Re-Do operation
* Known allergy to a pain medication in the protocol
* Existing contraindications to epidural catheter placement
* Requirement for 2 bars to be placed (rare)
* Inadequate baseline cognitive function to understand/respond to VAS questionnaire

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2006-10; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from patients undergoing pectus excavatum repair.
Pre-assignment Details: All patients who consented were enrolled
Groups:
- Epidural Group: Epidural analgesia arm of study
- PCA Group: IV narcotic analgesia arm of study
Period: Overall Study
Arm/Group | Epidural Group | PCA Group
Started | 55 (all enrolled completed) | 55 (all enrolled completed)
Completion of Study | 55 (all enrolled completed) | 55 (all enrolled completed)
Completed | 55 (all enrolled completed) | 55 (all enrolled completed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Group | PCA Group | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 53 | 102
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 15.3 (2.84) | 13.55 (2.91) | 14.43 (2.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 45 | 37 | 82
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Epidural Group | PCA Group
Number analyzed (Participants) | 55 | 55
days | 4.54 (1.01) | 4.25 (1.00)

2. Secondary Outcome: Time in the Operating Room
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Epidural Group | PCA Group
Number analyzed (Participants) | 55 | 55
hours | 1.97 (.35) | 1.58 (.33)

ADVERSE EVENTS:
Arm/Group | Epidural Group | PCA Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes